CLINICAL TRIAL: NCT02215031
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Intravenous Doses (10 to 50 mg) of BI 44370 BS Solution in Healthy Male Volunteers (Randomised, Single-blind, Placebo-controlled Within Dose Groups, Phase I)
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Rising Intravenous Doses of BI 44370 BS Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1246.12
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (2):
- BI 44370 (Experimental)
  Interventions: Drug: BI 44370
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 44370
  Arms: BI 44370
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to investigate safety, tolerability, and pharmacokinetics of BI 44370 BS solution for intravenous (i.v.) infusion

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR), Respiratory Rate (RR) and body temperature), 12-lead ECG, clinical laboratory tests
* Age 21 to 50 years inclusive
* Body Mass Index (BMI) 18.5 to 29.9 kg/m2 inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and German law

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR, RR, body temperature and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* Not willing to use adequate contraception (condom use plus another form of contraception, e.g. spermicide, oral contraceptive taken by female partner, sterilisation, or intrauterine device) during the whole study period from the time of the first intake of study drug until three months after the last intake

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant findings in vital signs | up to 16 days
Number of patients with clinically significant findings in 12-lead electrocardiogram (ECG) | up to 16 days
Number of patients with clinically significant laboratory findings | up to 16 days
Number of patients with adverse events | up to 37 days
Assessment of global tolerability by investigator on a 4-point scale | within 14 days after last trial procedure

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 24 hours after drug administration
tmax (time from dosing to maximum measured concentration) | up to 24 hours after drug administration
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after drug administration
%AUCtz-∞ (the percentage of the AUC0-∞ that is obtained by extrapolation) | up to 24 hours after drug administration
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 24 hours after drug administration
AUC0-2 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 2 hours after drug application) | up to 2 hours after drug administration
AUCt1-t2 (area under the concentration-time curve of the analyte in plasma over the time interval from time point t1 to time point t2) | up to 24 hours after drug administration
λz (terminal rate constant in plasma) | up to 24 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 24 hours after drug administration
MRTinf (mean residence time of the analyte in the body after intravenous administration) | up to 24 hours after drug administration
CL (total clearance of the analyte in plasma after intravascular administration) | up to 24 hours after drug administration
Vz (apparent volume of distribution during the terminal phase λz following an intravascular dose) | up to 24 hours after drug administration
Vss (apparent volume of distribution at steady state following intravascular administration) | up to 24 hours after drug administration
Aet1-t2 (amount of analyte eliminated in urine from the time point t1 to time point t2) | up to 24 hours after drug administration
fet1-t2 (fraction of analyte eliminated in urine from time point t1 to time point t2) | up to 24 hours after drug administration
CLR,t1-t2 (renal clearance of the analyte from the time point t1 until the time point t2) | up to 24 hours after drug administration